CLINICAL TRIAL: NCT01929252
Title: Phase 4 Study of Postoperative Analgesic Effect Of Dexmedetomidine Administration in Wound Infiltration For Total Abdominal Hysterectomy
Brief Title: Postoperative Analgesic Effect Of Dexmedetomidine Administration in Wound Infiltration for Total Abdominal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/07
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Pain
Keywords: dexmedetomidine; wound infiltration; postoperative analgesia
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator): %0.25 40 ml levobupivacaine and 2 mcg/kg dexmedetomidine administered via wound infiltration just before the incision.
  Interventions: Drug: Dexmedetomidine; Drug: Levobupivacaine
- Levobupivacaine (Active Comparator): %0.25 40 ml levobupivacaine administered via wound infiltration prior to incision.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — 2mcg.kg-1 dexmedetomidine wound infiltration
  Other Names: precedex
  Arms: Dexmedetomidine
Drug: Levobupivacaine — 0.25% levobupivacaine (40ml) wound infiltration
  Other Names: chirocaine

SUMMARY:
The aim of this study was to investigate the analgesic efficacy of dexmedetomidine administration in wound infiltration for total abdominal hysterectomy.

DETAILED DESCRIPTION:
Abdominal hysterectomy is associated with moderate to severe postoperative pain, effective analgesia after hysterectomy essential and several techniques are used such as administration of opioids, nonsteroidal anti-inflammatory drugs and wound infiltration of local anaesthetics. Different local anaesthetics can be used for the wound infiltration techniques.Ifiltration of the surgical wound with bupivacaine following outpatient provides pain relief in the postoperative period , allows the early discharge from the outpatient surgical units.There has been increased interest in administration of analgesic prior to surgical injury. Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with sedative , anxiolytic, analgesic, sympatholytic and antihypertensive effects.Dexmedetomidine has been used intravenously before initiation of anaesthesia and it has shown to provide some analgesic effect after surgery but there were some adverse hemodynamic effects. Surgical wound administration of dexmedetomidine may be useful to avoid the adverse haemodynamic effects of intravenous administration while still providing the postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yo female
* scheduled for elective hysterectomy
* no known allergies to drugs
* ASA 1=2 patients

Exclusion Criteria:

* history of diabetes
* history of chronic pain treatment
* pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Analgesic Consumption | 1 day after surgery
  Pethidine consumption (patient controlled analgesia procedure) was recorded

SECONDARY OUTCOMES:
Visual Analog Scale | 1 day after surgery
  Visual analog scale on rest and movement was recorded.
Haemodynamic Changes | During the surgery
  Arterial blood pressure, heart rate, peripheral oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Fatih M. Kurt, Resident, Principal Investigator — TC Erciyes University; Ayse Ulgey, Asst. Prof, Study Director — TC Erciyes University
Locations (1):
- Erciyes university hospital, Kayseri, Turkey (Türkiye)